CLINICAL TRIAL: NCT02138370
Title: Tissue Und Liquid Immune Biopsies to Predict Clinical Outcome in Localized Colorectal Cancer Patients - Retrospective Clinical Observational Study.
Brief Title: Comprehensive Immune-landscape in Localized Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: Immuno_CRC_001
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Colorectal Cancer; Immune Landscape
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- stage II and III colorectal cancer

SUMMARY:
Surgery still remains the mainstay of treatment for localized colorectal cancer. However, nearly 30% of patients with localized colorectal cancer (stage II and stage III) will present with recurrence. Tumor progression is mediated by both intrinsic genetic changes and by extrinsic epigenetic and host environmental factors, including interactions with the immune system. Several studies demonstrated that tumor infiltrating memory T-cells and type, density and location of infiltrating T cells are better predictors of disease-free survival in patients with CRC compared to the standard TNM staging. These data suggest that tumor invasion and progression are more accurately predicted by immune response in the primary tumor. In addition, mismatch repair (MMR)-deficient tumors are characterized a priori by a higher frequency of tumor infiltrating lymphocytes and are associated with significantly improved prognosis. Recently, Stotz et al showed that the preoperative lymphocyte to monocyte ratio in peripheral blood samples predicts clinical outcome in patients with stage III colon cancer. So far there is no comprehensive analysis of the immune-landscape in CRC.

The aim of the current project is to identify a comprehensive panel of immunomarkers in localized colorectal cancer (stage II and stage III) applicable for the detection of patients at high risk of recurrence. For the first time, specific tumor-infiltrating immune cells, mismatch repair protein expression in tumor tissue and preoperative blood based inflammatory markers from routine blood counts in corresponding peripheral blood samples and known clinicopathological features will be correlated with outcome in 300 localized CRC patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients ≥ 18 years of age;
* Formalin fixed paraffin embedded (FFPE) tissue samples of stage II and stage III colorectal cancer patients consecutively enrolled at the Division of Clinical Oncology, Department of Med.University of Graz (Graz, Austria) between 1995 - 2011

Exclusion Criteria:

* Male and Female patients < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with histopathologically confirmed stage II and III colon cancer consecutively enrolled at the Division of Clinical Oncology, Department of Medicine, Medical University of Graz (Graz, Austria) between 1995 and 2011.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Time to disease recurrence | 16 years

SECONDARY OUTCOMES:
overall survival | 16 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zuerich, Zurich, Canton of Zurich, Switzerland